CLINICAL TRIAL: NCT05381272
Title: Impact of Severe and Very Early Onset Intra-uterine Growth Restriction on Neurodevelopemental Outcome in Preterm Infants at 2 Years Old: a Monocentric Case Control Study
Brief Title: Impact of Early and Severe Fetal Growth Restriction on Neurodevelopmental Outcomes in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Apolline WITTWER, MD, Praticien Hospitalier, Central Hospital, Nancy, France
Other Study IDs: 2022PI010
Record Dates: First submitted 2022-04-13; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Severe Intra-uterine Growth Restriction; Preterm Birth; Neurodevelopmental Disorders; Placental Insufficiency
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders; Placental Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Infants born before 34 weeks of gestational age (WGA) with severe and early antenatal diagnosed intra uterine growth restriction
- Controls: infants born before 34 WGA at the same period, with no IUGR, apparied on sex and gestationnal age

SUMMARY:
Very early onset intra uterine growth restriction (IUGR) affects 5-10% of pregnancies and is the second leading cause of perinatal mortality.

However, there is few studies on this subject, especially concerning the neurodevelopment outcomes.

Objective: to compare neurodevelopmental outcomes at the age of 2 of very preterm infants with antenatal duagnosis of severe and early IUGR in comparison with infants of the same gestational age, same sex and over the same period with no IUGR.

Hypothesis : Preterm infants with early and severe antenatal IUGR have more neurodevelopmental delay than infants with no IUGR.

DETAILED DESCRIPTION:
Method: A monocentric retrospective case control study will be conducted at the Nancy University Hospital.

Each infant included (cases) will be match to 2 controls based on gestational age, period and sex which will allow us to individualize the impact of early and severe IUGR.

Inclusion criteria: Infants born before 34 weeks of gestational age, and whose antenatal files were discussed at the pluridisciplinary antenatal diagnosis center of Nancy from 2010 to 2020 with diagnosis of IUGR confirmed between 22 and 25 years of age. IUGR is defined by estimated fetal weight inferior to the 3rd percentile for the gestational age (calculated by the Hadlok formula and reported on the CFEF curves).

Exclusion criteria: Infants with anoxo ischemic encephalopathy or major neonatal surgery.

Cases and controls have a particular follow up thanks to the "Rafael" network which is a regional perinatal network following up preterm infants and infants at risk to have impairment in neurodevelopmental outcomes.

This follow up concerns general items and items based more specifically on neurodeveloppemental outcomes.

This neurodeveloppemental follow up at 2 years old is based on the ASQ scale witch explores 5 areas : communication, gross motor, fine motor, problem solving and personal social. Thanks to this follow up we will focus on the gross motor, social and communication.

The aim of the study is to analyze the different items of the neurodevelopment between the 2 groups. The hypothesis is that premature infants with severe and early growth restriction have a delay concerning psychomotor acquisitions.

Primary outcome: to compare neurodevelopmental outcomes at the age of 2 of very preterm infants with antenatal duagnosis of severe and early IUGR in comparison with infants of the same gestational age, same sex and over the same period with no IUGR (age of independant walking, gross motor, fine motor, communication, social items).

Secondary outcomes:

* complications during hospitalization between the 2 groups (incidence of necrotizing enterocolitis, early or late onset sepsis, retinopathy, intraventricular hemorrhage or abnormal MRI, audtion deficiency, bronchopulmonary dysplasia, persistent ductus arteriosus,...)
* neurodevelopment outcomes at 2 years of age
* growth (weight/height/CP) up to 2 years of age
* rehospitalizations during the first 2 years of life

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 34 weeks of gestational age, and whose antenatal files were discussed at the pluridisciplinary antenatal diagnosis center of Nancy from 2010 to 2020 with diagnosis of IUGR confirmed between 22 and 25 years of age. IUGR is defined by estimated fetal weight inferior to the 3rd percentile for the gestational age (Audipog curves).

Each infant included will be matched to 2 controls on gestational age, period and sex

Exclusion Criteria:

* no

Ages: 0 Days to 2 Years | Sex: All
Age Groups: Child
Study Population: Antenatal IUGR diagnosed preterm infants born before 34 weeks of gestational age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcomes at 2 years old evaluated by ASQ scale | at 2 years old
  This neurodeveloppemental follow up is based on the ASQ scale witch explores 5 areas : communication, gross motor, fine motor, problem solving and personal social.